CLINICAL TRIAL: NCT00170365
Title: Restorative Yoga for Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Hennepin Faculty Associates (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR-04-2412
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Stress; Anxiety
Keywords: Stress; Yoga
MeSH Terms: conditions — Anxiety Disorders

INTERVENTIONS:
Behavioral: Restorative Yoga

SUMMARY:
The study examined Restorative Yoga as a method of stress reduction for the HFA Addiction Medicine Clinic staff volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to determine if there is a perceived benefit from adding a restorative yoga class as a method of stress reduction for the HFA Addiction Medicine Clinic staff. Working in a busy clinic can be very stressful. While it is not always possible to completely eliminate stress from our lives, it is known that stress reduction techniques help to diminish the negative consequences of stress. This study was designed to answer the following question "How much change in perceived stress is obtained through weekly Restorative Yoga sessions?" Study population were members of the HFA Addiction Medicine Clinic. All staff completed the Spielberger Job Stress Survey and the State-Trait Anxiety Inventory at baseline and at six months following intervention onset. Volunteers from the Addiction Medicine Clinic attended weekly restorative yoga sessions 45 minutes in length held over the noon hour. Serial State-Trait Anxiety Inventory and weekly questionnaire regarding the perceived effects of the restorative yoga on aspects fo patient care were completed by study volunteers.

ELIGIBILITY:
Inclusion Criteria:

* member of HFA Addiction Medicine Clinic staff
* willing to participate in the restorative yoga sessions and to complete study instruments

Exclusion Criteria:

* unwilling to participate in the restorative ygoa sessions (assigned then to the control group)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2005-03

PRIMARY OUTCOMES:
The primary outcome measurement were the Spielberger State-Trait Anxiety Inventory scores.

SECONDARY OUTCOMES:
Secondary measurements were :
-number of sessions attended
-results of restorative yoga questionnaire on patient care and stress levels
-results of Job Stress Survey

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Wesa, M.D., Principal Investigator — Hennepin Faculty Associates/ Hennepin County Meical Center
Locations (1):
- Hennepin Faculty Associates/ Hennepin County Medica Center, Minneapolis, Minnesota, United States